CLINICAL TRIAL: NCT00311207
Title: Development of Tuberculosis Diagnostic Kit
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Taichung Veterans General Hospital (Other)
Other Study IDs: 940601/C05098
Record Dates: First submitted 2006-03-24; First posted 2006-04-05 (Estimated); Last update posted 2006-04-05 (Estimated); Status verified 2006-04

CONDITIONS: Tuberculosis; Lung Cancer; Pneumonia
Keywords: diagnostic kit; immunochromatography test; PCR detection kit; luminex
MeSH Terms: conditions — Tuberculosis; Lung Neoplasms; Pneumonia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other

SUMMARY:
Pulmonary tuberculosis is one of the most important infectious diseases in human with high mortality.

Early diagnosis followed by antibiotic treatment is the only way for control of the disease. However, most of commercial tuberculosis diagnostic kits are of moderate sensitivity. Oncoprobe Inc. recently developed a tuberculosis diagnostic kit (HR-103) based on detection of antibody against Mycobacterium tuberculosis in serum. The main purpose of this project is to evaluate the sensitivity and specificity of the kit in detection of pulmonary tuberculosis from saliva, urine, pleura and serum samples.Capilia TB assay and another Immunochromatographic assay such as ESAT-6 and CFP-10 based or other PCR based immunochromatographic assay will be tried to detection tuberculous disease.

DETAILED DESCRIPTION:
Sputum samples from 200 patients with chest or respiratory problems will be collected. Presence of M.

tuberculosis in the samples will be checked by acid-fast stain and bacterial culture and identification methods.

At the same time, saliva, urine, and serum samples from these 200 patients and 50 healthy volunteers will be collected. The tuberculosis diagnostic kit (HR-103) from Oncoprobe Inc. or capilia TB assay or another Immunochromatographic assay such as ESAT-6 and CFP-10 based or other PCR based immunochromatographic assay will be used to detect tuberculosis disease from these samples. By comparing the results with the stain and identification results of sputum samples from the 200 patients, the sensitivity and specificity of the kit in detection of pulmonary tuberculosis from saliva, urine,pleura and serum samples, as well as from combination of these samples, will be obtained. In addition to pulmonary tuberculosis, M. tuberculosis causes pleural tuberculosis. Diagnosis of pleural tuberculosis involves determination of activities of adenosine deaminase and interferon-gamma in pleural effusion, which is tedious. We also plan to collect pleural effusion samples from 100 patients, and examined by the tuberculosis diagnostic kit (HR-103) from Oncoprobe Inc. By comparing the results with the adenosine deaminase and interferon-gamma activities of the same samples, the sensitivity and specificity of the kit in detection of pleural tuberculosis from pleural effusion samples will be obtained.

ELIGIBILITY:
Inclusion Criteria: clinical suspicious of tuberculosis

-

Exclusion Criteria:

* HIV

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200
Dates: Start 2005-12; Study Completion 2006-11

CONTACTS AND LOCATIONS:
Overall Officials: Shen Gwan Han, MD, Principal Investigator — Respiratory and Critical care medicine department of Taichung Veterans General Hospital
Locations (1):
- Taichung Veterans General Hospital, Taichung, Taiwan